CLINICAL TRIAL: NCT01715623
Title: Polymorphism of the IgH Locus Regulatory Region as a Prognostic Factor During Immune Pathologies.
Acronym: PRIERR
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Direction Générale de la Santé, France (Other)
Responsible Party: Sponsor
Other Study IDs: I12002 PRIERR
Record Dates: First submitted 2012-10-22; First posted 2012-10-29 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers; Children With HSP; Subject With Allergy; Lymphoma
Keywords: polymorphism; serum Ig
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We previously showed that both antibody class switching (from IgM to IgG, IgA or IgE) and antibody secretion are controlled by a polymorphic "3' regulatory region" (3'RR) of the immunoglobulin heavy chain (IgH) locus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Children with HSP: children with Purpura of Henoch-Schönlein with or without renal complication
  Interventions: Biological: a blood sample
- healthy volunteers: healthy volunteers without allergy
  Interventions: Biological: a blood sample
- subjects with allergy: subjects with peanut allergy or hymenoptera venom allergy
  Interventions: Biological: a blood sample
- lymphoma: lymphoma-proliferation with chromosome 14 translocation
  Interventions: Biological: a blood sample

INTERVENTIONS:
Biological: a blood sample — Dosage of Ig

SUMMARY:
The investigators previously showed that both antibody class switching (from IgM to IgG, IgA or IgE) and antibody secretion are controlled by a polymorphic "3' regulatory region" (3'RR) of the immunoglobulin heavy chain (IgH) locus. Alleles of the 3'RR have shown influences on the severity and progression of IgA nephropathy (IgAN) (with an over-representation of the B allele among patients with severe kidney IgA deposits). Allele B also constitutes a risk factor for celiac disease, herpetiform dermatitis, psoriasis and rheumatoid arthritis. Since the 3'RR now appears as a crucial regulator of Ig production, we wish to check whether its genetic polymorphism might influence not only the occurrence of immunopathologic processes involving class-switched antibody deregulated production but also the severity of such diseases or the time course of their progression. We wish to focus on two conditions involving class-switched antibodies: on one hand the severe forms of IgE hypersensitivities, and on the other hand a disease involving pathogenic IgA and for which the prognosis is currently very difficult to predict at the onset of the disease: Henoch-Schonlein purpura (HSP).

Regarding hypersensitivities, the diversity of their clinical manifestations prompt us to focus on homogeneous groups of patients and we thus wish to concentrate on two groups of patients who are frequently referred to the hospital: severe allergies to Hymenoptera venoms and severe food allergies related to peanut allergens sensitization. These groups will be built by considering multiple clinical criteria (clinical history, severity of the manifestations, positive skin tests, and positive oral provocation tests for peanut allergens…) and biological criteria authenticating the mechanisms of the disease (high specific serum IgE, demonstration of specific basophil activation by the allergen…).

In parallel to the study in patients, we will include a large cohort of healthy controls (400 individuals), in order to be able to decipher whether correlations can be seen between:

* IgH 3'RR genotypes
* The serum accumulation of the various Ig classes, including IgG subclasses, IgA (which are sometimes depicted as protective, sometimes as tolerogenic and anti-inflammatory) and IgE (highly pro-inflammatory and responsible for hypersensitivities)
* IgG allotypes (with 6 frequent IgG haplotypes known in human and previously reported as correlated with varying levels of IgG and IgE production in normal individuals).

DETAILED DESCRIPTION:
This study should thus finally provide answers to 5 questions which are currently un-addressed:

* How the 3'RR alleles are linked to IgG allotypes and corresponding IgH haplotypes?
* Is there a physiological link between 3'RR alleles and production of the various Ig classes and sub-classes?
* Is the 3'RR polymorphism connected with the risk of more severe forms of allergic diseases?
* Is the 3'RR polymorphism connected with the risk of occurrence and/or severe evolution of HSP?
* Is the oncogenicity of translocations affecting the IgH locus connected to the strength of the 3'RR allelic variants?

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers:

Age ≥ 18 and < 50 years No history of allergy, haematological malignancies or immune diseases

* Subjects with allergy:
* Children:

Age ≥ 4 and < 18 years Clinical history supporting the diagnosis of severe food allergy Peanut specific IgE (Arah2) -Adults: Age > 18 and < 60 years History of severe reaction after antigenic challenge Anaphylactic shock already experienced Specific IgE or positive BAT Positive prick tests

* subject with HPS:
* Children:

Age ≥ 4 and < 18 years Henoch Schonlein Purpura (HSP) documented by Ankara 2008 criteria

-Adult: Henoch Schonlein Purpura(HSP) with renal involvement Adults ≥ 18 years,

Exclusion Criteria:

* subject with allergy or subject with Henoch Schonlein Purpura(HSP): known pregnancy patient under guardianship
* Healthy Volunteers:

Allergy known pregnancy patient under guardianship

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 4 populations :
  * Healthy Volunteers
  * subjects with HPS
  * subjects with peanut allergy or hymenoptera venom allergy
  * lymphoma (biological collection)
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
the percentage of allele B | one day
  A comparison will be made of the percentage of allele B between healthy volunteers and the three cohorts of subjects with various diseases: (1) lymphoma (lymphoma-proliferation with chromosome 14 translocation ), (2) Henoch-Schonlein purpura HSP (3), allergy (peanut and Hymenoptera venom)

CONTACTS AND LOCATIONS:
Overall Officials: Michel COGNE, MD, Principal Investigator — Limoges UH
Locations (4):
- France (4):
  - Clinical Investigation Center, Limoges
  - Nephrology, Limoges
  - Pediatric, Limoges
  - Pneumology, Limoges